CLINICAL TRIAL: NCT00674700
Title: A Randomized, DBPC, Multi-national Phase II/III Study of the Safety and Efficacy of Two Doses of Sublingual Immunotherapy (SLIT) Administered as Allergen-based Tablets Once Daily to Adult Patients Suffering From HDM Allergic Rhinitis
Brief Title: Safety and Efficacy Study of Sublingual Immunotherapy (SLIT) to Treat House Dust Mite Allergic Rhinitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Stallergenes Greer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VO57.07
Record Dates: First submitted 2008-05-06; First posted 2008-05-08 (Estimated); Results first posted 2016-05-19 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-04

CONDITIONS: Allergic Rhinitis
Keywords: House dust mites allergy
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Sublingual Immunotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 300 IR (Active Comparator): 300 IR house dust mites allergen extract tablet
  Interventions: Drug: 300 IR house dust mites allergen extract tablet
- 500 IR (Active Comparator): 500 IR house dust mites allergen extract tablet
  Interventions: Drug: 500 IR house dust mites allergen extract tablet
- Placebo (Placebo Comparator): Placebo tablet
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: 300 IR house dust mites allergen extract tablet — One sublingual tablet daily for one year
  Other Names: Sublingual immunotherapy tablet
  Arms: 300 IR
Drug: 500 IR house dust mites allergen extract tablet — One sublingual tablet daily for one year
  Other Names: Sublingual immunotherapy tablet
  Arms: 500 IR
Drug: Placebo tablet — One sublingual tablet daily for one year
  Other Names: Sublingual placebo tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy of two doses of sublingual immunotherapy (SLIT) administered as allergen-based tablets once daily over a period of 12 months compared to placebo, for reduction of allergic rhinitis symptoms and rescue medication usage

DETAILED DESCRIPTION:
Allergic rhinitis is a high-prevalence disease in many developed countries, affecting about 10 to 20% of the general population. House dust mite allergens are known to cause perennial allergic rhinitis.

In designing the present study, the guidelines proposed by the World Allergy Organization (WAO) task force for methodology of immunotherapy studies have been taken into consideration.

After a 2-month screening period, patients will be administered the dose of 300 IR- or 500 IR-house dust mite allergen-based tablets or placebo for a period of 12 months. The carry-over effect will be evaluated after a treatment-free follow up period of 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female outpatients aged 18 to 50 years (inclusive).
2. Patients who have been informed of the nature and aims of the study and have given their written consent
3. Patients must be in general good health as determined by past medical history, physical examination and safety laboratory tests.
4. Female patients of childbearing potential are eligible
5. Negative urine pregnancy test on female patients of childbearing potential.
6. House dust mite-related allergic rhinitis for at least 1 year.
7. Sensitised to D. pteronyssinus or D. farinae (positive SPT with wheal diameter greater than 3 mm and a specific IgE level ≥ 0.7 kU/L).
8. Baseline ARTSS > 5 (after completion of the 7-day daily record card).
9. Patients who are willing to comply with the protocol.
10. Patients who are able to understand the information given and the text of the consent form, and who are able to complete the daily record card and the RQLQ.

Exclusion Criteria:

1. Whatever the considered allergens, co-sensitisation leading to clinically relevant allergic rhinitis, sinusitis, conjunctivitis or asthma likely to significantly change the symptoms of the patient throughout the study (that means patient symptomatic to another allergen than house dust mites).
2. Patients with any nasal condition that could confound the efficacy or safety assessments (for example nasal polyposis).
3. Patients sensitised to cat or dog allergens and living with these animals at home.
4. Pregnant, breast-feeding / lactating or sexually active women of childbearing potential who are not using a medically accepted contraceptive method.
5. Asthma requiring treatment other than beta-2 inhaled agonists. Patients with intermittent asthma not necessitating inhaled or systemic corticoid treatment may be included (corresponding to the Global Initiative for Asthma [GINA] Step 1).
6. Patients treated with systemic, nasal or inhaled steroids (whatever the indication) within 4 weeks before Visit 1.
7. Patients treated with long acting systemic steroids (whatever the indication) within 12 weeks before Visit 1 and before Visit 2.
8. FEV1 < 80% of predicted value at Visit 1.
9. Patients who received allergy specific immunotherapy for house dust mites in the last 10 years.
10. Patients at risk of non-compliance.
11. Participation in any clinical study within the 12 weeks before Visit 1.
12. Investigators, co-investigators, as well as their children or spouses and all the study collaborators should not be enrolled in the study.
13. Any change in environmental measures for allergen avoidance during the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 509 (Actual)
Dates: Start 2007-10; Primary Completion 2009-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Christian BERGMANN, MD, Study Chair — Allergie-Centrum-Charité / ECARF

REFERENCES:
- [Result] Bergmann KC, Demoly P, Worm M, Fokkens WJ, Carrillo T, Tabar AI, Nguyen H, Montagut A, Zeldin RK. Efficacy and safety of sublingual tablets of house dust mite allergen extracts in adults with allergic rhinitis. J Allergy Clin Immunol. 2014 Jun;133(6):1608-14.e6. doi: 10.1016/j.jaci.2013.11.012. Epub 2013 Dec 31. PMID 24388010
- [Derived] Worm M, Demoly P, Okamoto Y, Vidal C, Daghildjian K, Yan K, Casale TB, Bergmann KC. Safety of 300IR house dust mite sublingual tablet from pooled clinical trial and post-marketing data. World Allergy Organ J. 2024 Jun 25;17(7):100924. doi: 10.1016/j.waojou.2024.100924. eCollection 2024 Jul. PMID 39035788
- [Derived] Baron-Bodo V, Batard T, Nguyen H, Frereux M, Horiot S, Harwanegg C, Bergmann KC, de Beaumont O, Moingeon P. Absence of IgE neosensitization in house dust mite allergic patients following sublingual immunotherapy. Clin Exp Allergy. 2012 Oct;42(10):1510-8. doi: 10.1111/j.1365-2222.2012.04044.x. PMID 22994348

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient First Visit 12 OCT 2007, Last Patient Last Visit 01 FEB 2010
Period: Year 1
Arm/Group | 300 IR | 500 IR | Placebo
Started | 170 | 169 | 170
Completed | 139 | 135 | 153
Not Completed | 31 | 34 | 17
Not completed — Adverse Event | 17 | 20 | 5
Not completed — Withdrawal by Subject | 7 | 7 | 6
Not completed — Any other reason not above-mentioned | 7 | 7 | 6
Period: Year 2 Follow-up Without Treatment
Arm/Group | 300 IR | 500 IR | Placebo
Started | 139 | 135 | 153
Completed | 133 | 123 | 141
Not Completed | 6 | 12 | 12
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 4
Not completed — Any other reason not above-mentioned | 5 | 10 | 7

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set included all participants who received at least one dose of the investigational product and had at least one Adjusted Symptom Score evaluation in the year.
Groups:
- Total: Total of all reporting groups
Arm/Group | 300 IR | 500 IR | Placebo | Total
Number analyzed (Participants) | 153 | 150 | 163 | 466
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.0 (8.52) | 30.1 (8.43) | 30.0 (8.96) | 29.7 (8.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 77 | 80 | 242
  Male | 68 | 73 | 83 | 224

OUTCOME MEASURES:

1. Primary Outcome: Average Adjusted Symptom Score (AAdSS) During the Year 1 Primary Period
Description: The AAdSS is derived from the daily Rhinoconjunctivitis Total Symptom Scores (RTSS), based on the severity of the 4 rhinitis symptoms: sneezing, rhinorrhoea, nasal pruritus and nasal congestion, each graded on a 4-point scale (0-3; 0: absent, 1: mild, 2: moderate, 3: severe).
  It ranges from 0 to 12, the higher the score the more severe the rhinitis.
Time Frame: Last 3 months of Year 1
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: Units on a scale (range: 0 to 12)
Arm/Group | 300 IR | 500 IR | Placebo
Number analyzed (Participants) | 141 | 136 | 153
Units on a scale (range: 0 to 12) | 3.18 (0.224) | 3.09 (0.230) | 3.87 (0.217)
Statistical Analysis 1: Comparison: 500 IR vs Placebo; Test type: Superiority or Other; p = 0.0066, ANCOVA — main effects = treatment and pools of study centers, Covariates = age, gender, asthma status, sensitization status and baseline ARTSS
Statistical Analysis 2: Comparison: 300 IR vs Placebo; Test type: Superiority or Other; p = 0.015, ANCOVA — main effects= treatment and pools of study centers, Covariates = age, gender, asthma status, sensitization status and baseline ARTSS

2. Secondary Outcome: Average Rhinitis Total Symptom Score (ARTSS)
Description: The Rhinitis Total Symptom Score (RTSS) evaluates the presence and severity of the 4 rhinitis symptoms: sneezing, rhinorrhoea, nasal pruritus and nasal congestion (absence of symptom (0), mild symptom (1), moderate symptom (2), severe symptom (3)). It ranges from 0 to 12, the higher the score the more severe the rhinitis.
Time Frame: Last 3 months of Year 1
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: Units on a scale (range: 0 to 12)
Arm/Group | 300 IR | 500 IR | Placebo
Number analyzed (Participants) | 141 | 136 | 153
Units on a scale (range: 0 to 12) | 2.74 (0.178) | 2.72 (0.183) | 3.32 (0.173)
Statistical Analysis 1: Comparison: 500 IR vs Placebo; Test type: Superiority or Other; p = 0.0086, ANCOVA
Statistical Analysis 2: Comparison: 300 IR vs Placebo; Test type: Superiority or Other; p = 0.0095, ANCOVA

ADVERSE EVENTS:
Time Frame: During the Year 1 with treatment and during the follow-up year without treatment. Results are provided here for the Year 1.
Description: Safety variables were adverse events (AEs) monitored throughout the study and data from physical examinations and clinical laboratory assessments.
Arm/Group | 300 IR | 500 IR | Placebo
Serious Adverse Events (participants affected / at risk) | 6/170 | 1/169 | 2/170
Other Adverse Events (participants affected / at risk) | 128/170 | 123/169 | 108/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 300 IR (N=170) | 500 IR (N=169) | Placebo (N=170)
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 — Reported as not related to the study drug.
Vaginal laceration (Reproductive system and breast disorders) | 1 | 0 | 0 — Reported as not related to the study drug.
Pharyngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Tubo-ovarian abscess (Infections and infestations) | 1 | 0 | 0 — Reported as not related to the study drug.
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 — Reported as not related to the study drug.
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 — Reported as not related to the study drug.
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 — Reported as not related to the study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 300 IR (N=170) | 500 IR (N=169) | Placebo (N=170)
Oral pruritus (Gastrointestinal disorders) | 51 | 43 | 8
Oedema mouth (Gastrointestinal disorders) | 21 | 28 | 1
Tongue oedema (Gastrointestinal disorders) | 9 | 10 | 1
Lip oedema (Gastrointestinal disorders) | 12 | 4 | 0
Nasopharyngitis (Infections and infestations) | 28 | 23 | 39
Influenza (Infections and infestations) | 15 | 14 | 16
Pharyngitis (Infections and infestations) | 17 | 10 | 19
Upper respiratory tract infection (Infections and infestations) | 11 | 5 | 9
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 42 | 36 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 16 | 18
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 6 | 11 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 10 | 10
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 7 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 2 | 6
Headache (Nervous system disorders) | 23 | 24 | 33
Eczema (Skin and subcutaneous tissue disorders) | 4 | 3 | 9
Ear pruritus (Ear and labyrinth disorders) | 4 | 13 | 1
Pyrexia (General disorders) | 4 | 1 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No